CLINICAL TRIAL: NCT06195930
Title: A Phase 2b Open-label Clinical Study to Evaluate the Tolerability and Safety of an Initiation Dose of 5 mg of Vericiguat in Participants With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: A Study to Learn How Safe Starting Vericiguat at a Dose of 5 Milligrams is in Participants With Chronic Heart Failure With Reduced Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21683; 2023-507682-25-00 (Other: CTIS)
Record Dates: First submitted 2023-12-07; First posted 2024-01-08 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: This is a multi-center, single arm, open label study of vericiguat initiation at 5 mg in HFrEF patients with EF <45%. The total study duration is approximately 4 weeks, including a 2-week screening period and a 2-week treatment period .
  Screening: Approximately 120 participants will be screened to achieve at least 100 participants who are assigned to study intervention and complete the treatment period of up to 2 weeks. Participants will undergo a screening visit to assess eligibility. Eligible participants must wait a mandatory 2 weeks before returning for Visit 1 in order to be clinically and hemodynamically stable.
  Treatment: At Visit 1, participants will receive vericiguat 5 mg (on top of standard of care) with directions to take once daily for 2 weeks. Participants will return for a study visit (Visit 2) after 2 weeks of treatment.
  Unscheduled visits may be utilized between Visits 1 and 2 at the discretion of the investigator for AE review and reporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Overall study (Experimental): At Visit 1 participants will receive 1x 5 mg Vericiguat (BAY1021189) tablet daily (on top of standard of care) for at least 14 days to max 18 days (+4 days time window allowed)
  Interventions: Drug: Vericiguat (BAY1021189) 5 mg

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) 5 mg — Vericiguat (BAY1021189) will be taken as 5 mg tablet 1x daily over at least 14 days up to 18 days (+ 4 days time window allowed)

SUMMARY:
Researchers are looking for a better way to treat people who have chronic heart failure with reduced ejection fraction. Chronic heart failure with reduced ejection fraction (HFrEF) is a long-term condition that occurs when the heart is too weak to pump enough blood to the rest of the body. This results in a reduced supply of the oxygen that the body requires to function properly. The common symptoms of HFrEF include breathlessness, weakness, fatigue, and swelling in the ankles and legs. If left untreated, heart failure can lead to other serious health problems, including damage to other organs, which may result in hospital stays or even death.

Vericiguat is an approved drug for use in people with chronic HFrEF. It works by activating a protein called soluble guanylate cyclase, which helps dilating the blood vessels and in turn improves heart function.

Currently, treatment with vericiguat starts at a daily dose of 2.5 milligrams (mg), which increases to 5 mg after 2 weeks. The dose is then increased to the target dose of 10 mg after another 2 weeks.

In this study, researchers are trying to learn how well participants can tolerate and how safe it is to start vericiguat at a dose of 5 mg. Starting directly at the 5 mg dose is expected to help reach the target dose of 10 mg faster. Participants will take vericiguat 5 mg as a tablet by mouth once daily along with their regular heart medications.

At the start of the study, study doctors will check participants' medical history and perform full health check-ups to confirm if they can take part in the study. Throughout the study, study doctors will monitor participants' previous and current medications, their heart health, and their overall well-being. This will help researchers assess how safe the study drug is and if they experience adverse events. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective of whether they think they are related to the study treatment.

Access to study treatment after the end of this study is not planned. Everyone, including study doctors and participants, will know what drug the participants receive during the study. Participants may be in the study for about 4 weeks.

Participants may not benefit from the treatment as the study is designed to assess safety and tolerability: the duration of the study is very short and participants will be taking a low dose of vericiguat without moving to the target dose of 10 mg during the study. However, the findings of this study may enable people with chronic HFrEF to safely skip one initial dosing step and reach the target dose of vericiguat faster.

Participants may experience medical problems such as low blood pressure, upset stomach, nausea, dizziness, and headache. Researchers will monitor and manage all these, and other, medical problems participants may have during the study.

ELIGIBILITY:
Inclusion Criteria:

* Has an Left ventricle ejection fraction (LVEF) of <45% assessed within 12 months before Visit 1 by local any imaging method, and no subsequent LVEF measurement > 45%. The most recent measurement must be used to determine eligibility.
* systolic blood pressure (SBP) ≥ 100 mmHg at screening and Visit 1 (pre-treatment).
* No changes in guideline-directed medical therapy for heart failure (GDMT) dosing (including beta blockers, angiotensin-converting enzyme inhibitor/ angiotensin II receptor blocker (ACEI/ARBs), angiotensin receptor-neprilysin inhibitor (ARNI), mineralocorticoid receptor antagonist (MRAs), hydralazine-nitrate combinations, sodium-glucose cotransporter 2 i(SGLT2) inhibitors, ivabradine, or oral diuretics):

  * Within 4 weeks of screening for participants without a heart failure (HF) event ≤6 months prior to screening
  * within 2 weeks of screening for participants with a HF event ≤6 months prior to screening
  * planned during study participation
* No expected medical procedures to occur 2 weeks before screening or during study participation.
* Participants with ( group 1) OR without (group 2) recent worsening HF event Group 1: History of chronic HF (NYHA class II symptomatic-IV) on GDMT with recent HFevent within 6 months of screening or outpatient IV / SC diuretic use within 3 months before screening.

OR Group 2: History of chronic HF (NYHA class II symptomatic-IV) on GDMT without recent HF event within 6 months of screening or outpatient intravenous/ subcutaneous (IV / SC) diuretic use within 3 months before screening.

Exclusion Criteria:

* History of symptomatic hypotension 4 weeks before screening
* Primary valvular heart disease requiring surgical procedure or intervention or has undergone a vascular surgical procedure or intervention within 3months before visit 1
* Hypertrophic cardiomyopathy
* Acute myocarditis or Takotsubo cardiomyopathy
* Awaiting heart transplantation (United Network for Organ Sharing Class 1A /1B or equivalent) or has or anticipates receiving an implanted ventricular assist device, or has received a heart transplant.
* Tachycardia-induced cardiomyopathy and/or uncontrolled tachyarrhythmia.
* Acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction (NSTEMI), or ST elevation myocardial infarction (STEMI), undergone coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within 3months before Visit 1, or indication for coronary revascularization at the time of treatment assignment.
* Symptomatic carotid stenosis, transient ischemic attack (TIA), or stroke within 3 months before Visit 1.
* History of repaired or unrepaired simple congenital heart disease (e.g., atrial or ventricular septal defects, or patent ductus arteriosus) with ongoing hemodynamically significant residual lesions, or any history of complex congenital heart disease (e.g. tetralogy of Fallot, transposition of the great arteries, single ventricle disease) regardless of repair status.
* Active endocarditis or constrictive pericarditis.
* Hemodynamic instability or hypovolemia within 4 weeks of screening and during the screening period.
* Currently hospitalized.
* estimated glomerular filtration rate (eGFR) based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation of <15 mL/min/1.73 m2 within 30 days before Visit 1 or on chronic dialysis. For participants with multiple eGFR results during screening, the most recent value will be used to determine eligibility.
* Severe hepatic insufficiency defined as albumin to bilirubin ratio (ALBI) Grade 3 or hepatic encephalopathy, or has hepatic laboratory abnormalities (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 ×upper limit of normal (ULN) or total bilirubin ≥2 × ULN). Exceptions for Gilbert's syndrome will be considered. Albumin, ALT, AST, and total bilirubin results within 30 days before Visit 1 may be used for assessment of laboratory abnormalities or the calculation of the ALBI score. For participants with multiple albumin and/or total bilirubin results during screening, the most recent value for each test will be used to calculate ALBI score.
* Malignancy or other noncardiac condition limiting life expectancy to <3years.
* Requires continuous home oxygen for severe pulmonary disease.
* Interstitial lung disease.
* Known allergy or hypersensitivity to vericiguat, any of its constituents, or any other soluble guanylate cyclase (sGC) stimulator.
* Amyloidosis or sarcoidosis.
* Concurrent or anticipated concomitant use of phosphodiesterase type 5 (PDE5) inhibitors such as vardenafil, tadalafil, and sildenafil during the study.
* Concurrent use of an sGC stimulator such as riociguat or vericiguat.
* Prior (within 2 weeks prior to screening) or anticipated concomitant administration of IV / SC diuretics or inotropes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (5):
  - Advanced Cardiovascular, LLC - Alexander City, Alexander City, Alabama
  - Reid Physician Associates | Cardiology Department, Richmond, Indiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - St. Louis Heart & Vascular, PC, St Louis, Missouri
  - Chear Center LLC, New York, New York
- Argentina (5):
  - Centro de Investigacion y Prevencion Cardiovascular | Sede Recoleta, Buenos Aires, Ciudad Auton. de Buenos Aires
  - CEDIC Centro de Investigación Clínica | Buenos Aires, Argentina, CABA, Ciudad Auton. de Buenos Aires
  - Consultorios Integrados Rosario | Instituto Medico de la Fundacion de Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto de Cardiologia de Corrientes Juana F. Cabral | Corrientes, Argentina, Corrientes
  - Centro de Investigaciones Clinicas del Litoral | Santa Fe, Argentina, Santa Fe
- Hungary (6):
  - Semmelweis Egyetem Belgyógyaszati és Haematológiai Klinika, Kardiológia, Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Coromed Smo Kft, Pécs
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
  - Complex Rendelo Med Zrt., Székesfehérvár
- Italy (4):
  - ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - IRCCS Centro Cardiologico Monzino, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
- Poland (7):
  - Malopolskie Centrum Sercowo-Naczyniowe PAKS, Chrzanów
  - Vita Longa Sp. z o.o., Katowice
  - Centrum Medyczne Zdrowa, Krakow
  - Clinical Best Solutions Sp. Z O.O. Sp.K., Lublin
  - NZOZ "Twoja Przychodnia" Sp. z o.o., Lublin
  - IRMED Osrodek Badan Klinicznych, Piotrkow Trybunalski
  - Clinical Best Solutions Sp. Z O.O. Sp.K., Warsaw
- Spain (6):
  - Hospital Clinico Universitario de Santiago de Compostela | Cardiology Department, Santiago de Compostela, A Coruña
  - Hospital del Mar | Cardiology Department, Barcelona
  - Hospital Universitari de Bellvitge | Bellvitge Biomedical Research Institute - Cardiology Department, Barcelona
  - Hospital Ramon y Cajal | Cardiology - Research Unit, Madrid
  - Hospital la Paz, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- Sweden (2):
  - Capio Citykliniken - Hjartmottagning, Lund
  - Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the NCT number or Bayer Study ID in the search field. — https://clinicaltrials.bayer.com/study/21683

RESULTS

PARTICIPANT FLOW:
Groups:
- Vericiguat 5 mg: Participants who started with study intervention intake: Vericiguat 5 mg - At Visit 1, subjects received vericiguat (BAY1021189) 5 mg oral as tablet (on top of standard of care) with directions to take once daily for 14 days (up to 18 days: +4 day time window allowed).
Period: Overall Study
Arm/Group | Vericiguat 5 mg
Started (Started Treatment Phase) | 106 (All participants in this study received Vericiguat 5 mg)
Participants With Worsening Heart Failure (HF) (Part of Vericiguat 5mg group: Participants who started study treatment with recent worsening Heart failure (HF) event) | 53 (Sub-group of the overall vericiguat 5 mg group to better differentiate the outcome measures.)
Participants Without Worsening Heart Failure (HF) (Part of Vericiguat 5mg group: Participants who started study treatment without recent worsening Heart failure (HF) event) | 53 (Sub-group of the overall vericiguat 5 mg group to better differentiate the outcome measures.)
Completed (Completed Treatment Phase) | 102
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Vericiguat 5 mg
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participant Age distribution
  Years | 66.9 (11.3)
Age, Customized [Count of Participants; unit: Participants] — Age Classification Type 1: Adults (between 18 and 64 years); From 65 to 84 years; 85 years and over
  Participants
    between 18 and 64 years | 42
    from 65 to 84 years | 61
    85 years and over | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Participant Disposition
  Participants
    Female | 30
    Male | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 102
  More than one race | 0
  Unknown or Not Reported | 1
History of HF event [Count of Participants; unit: Participants] — Participants with recent worsening Heart failure (HF) event (Group 1), Participants without recent worsening HF event (Group 2)
  Participants
    Participants with recent worsening HF event (Group 1) | 53
    Participants without recent worsening HF event (Group 2) | 53

OUTCOME MEASURES:

1. Primary Outcome: Treatment Tolerability: Number of Participants Without Discontinuation of Study Intervention (Incl. Max. 1 Day Interruption) and Without Moderate to Severe Symptomatic Hypotension
Description: Treatment tolerability, defined as the completion of the two-week 5 mg dose without discontinuation of study intervention (incl. max. 1 day interruption) and without moderate to severe symptomatic hypotension between Visit 1 and Visit 2
Time Frame: Between Visit 1 (Day 1) and Visit 2 (Day 14 up to Day 18 if +4 days time window is used)
Population: Safety Analysis Set (SAF) = 106 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vericiguat 5 mg
Number analyzed (Participants) | 106
Participants | 99

2. Secondary Outcome: Number of Participants With Any Adverse Event (AE) Reported Between Visit 1 and Visit 2
Description: Any AE reported between Visit 1 and Visit 2 to describe the safety events of initiation of 5mg dose.
Time Frame: Between Visit 1 (Day 1) and Visit 2 (Day 14 up to Day 18 if +4 days time window is used)
Population: Safety Analysis Set (SAF) = 106 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vericiguat 5 mg
Number analyzed (Participants) | 106
Participants | 14

3. Secondary Outcome: Number of Participants With no AE Related to Study Intervention Between Visit 1 and Visit 2
Description: Absence of AEs related to study intervention between Visit 1 and Visit 2 to describe safety events of initiation of 5mg dose.
Time Frame: Between Visit 1 (Day 1) and Visit 2 (Day 14 up to Day 18 if +4 days time window is used)
Population: Safety Analysis Set (SAF) = 106 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vericiguat 5 mg
Number analyzed (Participants) | 106
Participants | 96

4. Secondary Outcome: Number of Participants With Continuous Intake of Study Intervention Between Visit 1 and Visit 2 or Restart of Study Intervention After Any Temporary Interruption.
Description: To further evaluate the tolerability of 5mg as a starting dose
Time Frame: Between Visit 1 (Day 1) and Visit 2 (Day 14 up to Day 18 if +4 days time window is used)
Population: Safety Analysis Set (SAF) = 106 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vericiguat 5 mg
Number analyzed (Participants) | 106
Participants | 102

5. Primary Outcome: Treatment Tolerability: Number of Participants Without Discontinuation of Study Intervention (Max. 2 Day Interruption Included) and Without Moderate to Severe Symptomatic Hypotension
Description: Treatment tolerability, defined as the completion of the two-week 5 mg dose without discontinuation of study intervention (incl. max. 2 day interruption) and without moderate to severe symptomatic hypotension between Visit 1 and Visit 2
Time Frame: Between Visit 1 (Day 1) and Visit 2 (Day 14 up to Day 18 if +4 days time window is used)
Population: Safety Analysis Set (SAF) = 106 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vericiguat 5 mg
Number analyzed (Participants) | 106
Participants | 102

ADVERSE EVENTS:
Time Frame: Between Visit 1 (Day 1) and Visit 2 (Day 14 up to Day 18 if +4 days time window is used)
Arm/Group | Vericiguat 5 mg
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 1/106
Other Adverse Events (participants affected / at risk) | 14/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat 5 mg (N=106)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat 5 mg (N=106)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 7 (10)

LIMITATIONS AND CAVEATS:
Study Design: This analysis is based on a single-arm design, which may limit the generalizability of the findings. The absence of a control group restricts our ability to make definitive conclusions about the tolerability and safety of starting vericiguat at 5 mg/day to standard care or placebo. The results are based on descriptive statistics, which provide a summary of the data but do not infer causality or generalizability to a broader population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CONSULTANT agrees that it will nit use the Confidential Information, which consultant is required hereunder to keep confidential, for any purposes other than the provision of services, without first entering into a written agreement signed by the consultant and Bayer covering the use thereof.

DOCUMENTS (2):
  • Study Protocol (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT06195930/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT06195930/SAP_001.pdf